CLINICAL TRIAL: NCT06457412
Title: Programme for Intervention in Paediatric Obesity
Acronym: PinPo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Universidad de Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PinPo
Record Dates: First submitted 2024-05-27; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Childhood
Keywords: Obesity; Childhood; Grupal intervention
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Intervention group for the treatment of childhood obesity
  Interventions: Other: Intervention group for the treatment of childhood obesity

INTERVENTIONS:
Other: Intervention group for the treatment of childhood obesity — Intervention for children aged 6 to 12 years with childhood obesity (with a BMI greater than the 99th percentile), fostering motivation and encouraging changes toward healthy lifestyle habits to achieve greater adherence and to improve health. The program comprises 9 educational sessions designed by specialized professionals (code of Spanish register: 2007144741729) to be conducted in a health center. The sessions will be held every 15 days, with a duration of 90 minutes for a group of 10 children and another group of 10 family members and/or caregivers. Professionals from different disciplines (paediatricians, psychologists, nurses and nutritionists), will meet with groups of pediatric patients and in another group with their family members or primary caregivers.

SUMMARY:
The PinPo program aims to carry out a comprehensive intervention for children aged 6 to 12 years with childhood obesity (with a BMI greater than the 99th percentile), fostering motivation and encouraging changes toward healthy lifestyle habits to achieve greater adherence and improved health. The program comprises 9 educational sessions designed by specialized professionals from various disciplines (pediatrics, psychology, nursing, nutrition), for a group of 10 children and another group of 10 family members and/or caregivers. These sessions are conducted in a hospital setting every 15 days, each lasting 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 12 years old, with a BMI greater than the 99th percentile according to Cole criteria (2004).

Exclusion Criteria:

* Children < 6, or > 12 years.
* Children with chronic diseases or following a therapeutic diet.
* Children with intervention in other centers.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | 4 months
  The daily energy intake will be estimated using data from three internationally validated questionnaires: the adapted Consumption Frequency Questionnaire (CFC), the NHANES Food Questionnaire, and the Kidmed Test. The unit of measurement is kilocalories.
Diet composition | 4 months
  The composition of the diet by macronutrients and micronutrients will be estimated using data from three internationally validated questionnaires: the adapted Consumption Frequency Questionnaire (CFC), the NHANES Food Questionnaire, and the Kidmed Test. The unit of measurement is grams.

SECONDARY OUTCOMES:
Physical activity and sedentary behavior | 4 months
  Physical activity and sedentary behavior will be assessed in terms of time using an ad hoc questionnaire. The unit of measurement is minutes.
Screen Time | 4 months
  Screen time (including television, computers, cell phones, video games, and consoles) will be assessed in terms of time using an ad hoc questionnaire. The unit of measurement is minutes of screen display.
Height | 4 months
  Height in centimeters is measured with the SECA 213 precision measuring instrument.
Weight | 4 months
  Weight in grams is measured by the precision weighing scale model Tanita 780PMA
Body mass index | 4 months
  Body mass index in kilograms per square meter is calculated.
Waist circumference | 4 months
  Waist circumference in centimeters is measured with a CESCORF measuring tape
Self-esteem | 4 months
  Self-esteem will be evaluated using ad hoc questionnaires. It will be measured by obtaining a score.
Confidence | 4 months
  Confidence will be evaluated using ad hoc questionnaires. It will be measured by obtaining a score.
Emotional Regulation | 4 months
  Emotional regulation will be evaluated using ad hoc questionnaires. It will be measured by obtaining a score.
Hematological analysis: Hemoglobine | 4 months
  Hemoglobin levels are determined in grams per deciliter on an individual basis.
Hematological analysis: Hematocrite | 4 months
  Hematocrite levels are determined in percentage on an individual basis.
Hematological analysis: Erythrocytes | 4 months
  Erythrocytes count is measured in 10e06 units per microliter on an individual basis.
Hematological analysis: Mean corpuscular volume | 4 months
  Mean corpuscular volume is measured in femtoliters on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin | 4 months
  Mean corpuscular hemoglobine is measured in picograms on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin concentration | 4 months
  Mean corpuscular hemoglobine concentration is measured in grams per deciliter on an individual basis.
Hematological analysis: Red cell blood distribution width | 4 months
  Red cell blood distribution width is determined in percentage on an individual basis.
Hematological analysis: White blood cells | 4 months
  White blood cells count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Neutrophils | 4 months
  Neutrophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Lymphocytes | 4 months
  Lymphocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Monocytes | 4 months
  Monocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Eosinophils | 4 months
  Eosinophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Basophiles | 4 months
  Basophiles count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Platelets | 4 months
  Platelets count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Mean platelet volume | 4 months
  Mean platelet volume is measured in femtoliters on an individual basis.
Biochemical analysis: Glucose | 4 months
  Glucose is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Bilirubin | 4 months
  Total bilirubin is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma
Biochemical analysis: Creatinine | 4 months
  Creatinine is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urate | 4 months
  Urate is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urea | 4 months
  Urea is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total protein | 4 months
  Total protein is measured both in grams per deciliter and in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Aspartate aminotransferase | 4 months
  Aspartate aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alanine aminotransferase | 4 months
  Alanine aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Gamma-glutamyl transferase | 4 months
  Gamma-glutamyl transferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alkaline phosphatase | 4 months
  Alkaline phosphatase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total cholesterol | 4 months
  Total cholesterol is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: High density lipoproteins | 4 months
  High density lipoproteins (HDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Non-HDL cholesterol | 4 months
  Non-HDL cholesterol levels are calculated in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Low density lipoproteins | 4 months
  Low density lipoproteins (LDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein A1 | 4 months
  Apolipoprotein A1 is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein B | 4 months
  Apolipoprotein B is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Calcium | 4 months
  Calcium is measured both in milligrams per deciliter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Potassium | 4 months
  Potassium is measured both in millimoles per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sodium | 4 months
  Sodium is measured in millimoles per liter, in milliequivalents per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Phosphorus | 4 months
  Phosphorus is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Iron | 4 months
  Iron is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Magnesium | 4 months
  Magnesium is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Zinc | 4 months
  Zinc is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin | 4 months
  Insulin is measured both in micro international units per liter and in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin resistance | 4 months
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) index is used to estimate insulin resistance.
Biochemical analysis: C-reactive protein | 4 months
  C-reactive protein is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Tumor necrosis factor alpha | 4 months
  Tumor necrosis factor alpha is measured in picograms per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Adiponectin | 4 months
  Adiponectin is measured in milligrams per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Energy | 4 months
  Adiponectin is measured in milligrams per liter on an individual basis. Analysis performed Energy is determined in kilocalories on an individual basis. Analysis performed in plasma.
Biochemical analysis: Carbohydrates | 4 months
  Adiponectin is measured in milligrams per liter on an individual basis. Analysis performed Carbohydrates are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sugars | 4 months
  Sugars are measured in grams on an individual basis. Analysis performed in plasma.Carbohydrates are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Fiber | 4 months
  Fibers are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polysaccharides | 4 months
  Polysaccharides are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total fat | 4 months
  Total fat is measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Saturated fatty acids | 4 months
  Saturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Monounsaturated fatty acids | 4 months
  Monounsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polyunsaturated fatty acids | 4 months
  Polyunsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B1 | 4 months
  Vitamin B1 is measured in milligrams on an individual basis. Analysis performed in plasma
Biochemical analysis: Vitamin B2 | 4 months
  Vitamin B2 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B3 | 4 months
  Vitamin B3 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B6 | 4 months
  Vitamin B6 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B9 | 4 months
  Vitamin B9 is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B12 | 4 months
  Vitamin B12 is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin C | 4 months
  Vitamin C is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin A | 4 months
  Vitamin A is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin D | 4 months
  Vitamin D is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin E | 4 months
  Vitamin E is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Carotenes | 4 months
  Carotenes are measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Retinol | 4 months
  Retinol is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Water | 4 months
  Water is measured in grams on an individual basis. Analysis performed in plasma.
Fecal microbiome: DNA | 4 months
  Samples will be homogenized in a Stomacher-400 blender. Subsequently, a QIAamp DNA Stool Mini Kit (QIAGEN, Barcelona, Spain) will be used for the DNA extraction as indicated by the manufacturer with the exception of the incubation at 70 °C, since the samples will be mixed with the lysis buffer and incubated at a temperature of 95 °C to ensure that both Gram-positive and Gram-negative bacteria are lysed. The quantification of the DNA will be conducted with a NanoDrop ND1000 spectrophotometer (Thermo Fisher Scientific, DE, USA) and the DNA yield will be calculated by measuring absorbance ratios spectrophotometrically, including A260/230 nm for salt and phenol contamination and A260/280 nm for protein contamination. The unit of measurement is percentage of abundance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No